CLINICAL TRIAL: NCT05259358
Title: The Effect of Muscular Endurance on Disability Level and Participation in Life in Non-specific Neck Pain
Brief Title: The Effect of Muscular Endurance on Disability Level and Participation in Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Burcu Özüberk, Principal Investigator, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72867572-050.01.04-95509
Record Dates: First submitted 2022-01-15; First posted 2022-02-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain
Keywords: non specific neck pain; endurance; disability; participation; pain
MeSH Terms: conditions — Neck Pain; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients included in the treatment group had 10 sessions postural smoothness, Chin tuck exercises, Range of motion exercises at all angles of the cervical joint, Neck isometric exercises, Cervical stabilization exercises (with ball), Pectoralis, latissimus dorsi, trapezoidal upper part, rhomboid and scalene muscle stretching exercises will be done face-to-face with a physiotherapist. At the end of 10 sessions of face-to-face training, the patients will perform the same exercises at home for 1 month. The patients will not given any exercises in the control group. Measurements and evaluations of the patients in both groups will be made twice that is before and after the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Active Comparator): In addition to routine treatment:
  Postural evenness
  Chin tuck exercise
  Range of motion exercises for all angles of the cervical joint
  Neck isometric exercises
  Cervical stabilization exercises (with ball)
  Stretching exercises of pectoralis, latissimus dorsi, trapezius upper part, levator scapula, rhomboid and scalene muscles
  Interventions: Other: exercise
- routine (No Intervention): only routine treatment

INTERVENTIONS:
Other: exercise — exercises that increase muscular endurance
  Arms: exercise

SUMMARY:
Non-specific neck pain (NSBA), which is one of the most common causes of neck pain in the literature, occurs as a result of a postural or mechanical cause without a specific pathology or injury to the musculoskeletal system. NSBA causes an increase in superficial cervical muscle activity, and a decrease in deep cervical muscle activity, which contains a large amount of muscle spindles. Patients with chronic neck pain face functional limitations in many ways. Evaluation of disability as a result of loss of functions related to neck pain is necessary to cope with neck pain. In the ICF activity and participation section due to neck pain, it is stated that the daily life activities of the person are limited due to neck pain, both at work and at home, and with this, the level of disability of the person increases. Loss of endurance, on the other hand, appears as a physical marker in the development of chronic neck pain due to the effect of muscle functions in patients who have problems in the neck region, according to ICF.

DETAILED DESCRIPTION:
Patients with non-specific neck pain who volunteered to participate in the study and who met the inclusion criteria of the study will be included in the study after signing the voluntary consent form. First of all, the demographic and clinical characteristics of the patients will be questioned with the evaluation form. The personal information of the patients (gender, height, weight, smoking, etc.) and clinical status (pain type, pain intensity, muscle endurance measurements) will be recorded by the physiotherapist in the evaluation form. In addition to the evaluation form, the Northwick Park Neck Pain Questionnaire will evaluate the patients' neck disability, while the Keele Participation Evaluation will evaluate their level of participation in life.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent to participate in the study
* Clinical diagnosis of non spesific neck pain

Exclusion Criteria:

* There is physical/mental problem that may prevent exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
KEELE ASSESMENT OF PARTICIPATION | change in participation in life in one month
  participation in life: 15 items total; min:0; max:11; 1-11:participation restriction in at least
  one activity. Mobility; Self-Care; Domestic Life; Interpersonal Interactions and Relationships; Major Life Areas; Community Social & Civic life
  Mean response for each question was reported, with a lower score indicating better perceived participation; question scores range from 1 to 5
Northwick Park Neck Pain Questionnaire | change in disability level in one month
  the neck pain and the consequent patient disabilities: The neck pain score is the sum of the points scored for the first nine questions.
  Question 9 (about the driving) is not applicable if the patient doesn't drive a car in good health.
  • If the nine questions are answered: NPQ percentage = ((neck pain score) / 36) x 100%.
  • If the first eight questions are answered: NPQ percentage = ((neck pain score) / 32) x 100%. The higher the percentage, the greater the disability and the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mine A Deniz, PT, PhD, Study Director — Suleyman Demirel University
Locations (2):
- Turkey (Türkiye) (2):
  - Suleyman Demirel University Education and Training Hospital, Isparta, East Campus
  - Suleyman Demirel University, Isparta, East Campus